CLINICAL TRIAL: NCT03478969
Title: Patient-Reported Outcomes With the Accu-Chek® Solo Micropump System vs. Multiple Daily Injection Therapy vs. Mylife OmniPod® in Patients With Type 1 Diabetes
Brief Title: Participant-Reported Outcomes With the Accu-Chek® Solo Micropump System
Acronym: PRO Solo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD002718
Record Dates: First submitted 2018-03-13; First posted 2018-03-27 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Accu-Chek® Solo (Experimental): Continuous subcutaneous insulin infusion (CSII) with Accu-Chek® Solo Micropump system for 26 weeks. From Week 26 until Week 39, all Groups will be using the Accu-Chek® Solo Micropump system for CSII therapy.
  Interventions: Device: Accu-Chek® Solo micropump system
- Group B: MDI, then Accu-Chek® Solo (Experimental): Multiple daily injections (MDI) for 26 weeks. From Week 26 until Week 39, all Groups will be using the Accu-Chek® Solo Micropump system for CSII therapy.
  Interventions: Device: Accu-Chek® Solo micropump system; Other: Multiple Daily Injections (MDI) therapy
- Group C: mylife™ OmniPod®, then Accu-Chek® Solo (Experimental): Continuous subcutaneous insulin infusion (CSII) with the mylife™ OmniPod® Insulin Management system for 26 weeks. From Week 26 until Week 39, all Groups will be using the Accu-Chek® Solo Micropump system for CSII therapy.
  Interventions: Device: Accu-Chek® Solo micropump system; Device: mylife™ OmniPod® Insulin Management System

INTERVENTIONS:
Device: Accu-Chek® Solo micropump system — Medical device for subcutaneous delivery of insulin in a personalized way.
Device: mylife™ OmniPod® Insulin Management System — A patch pump system delivering insulin.
  Arms: Group C: mylife™ OmniPod®, then Accu-Chek® Solo
Other: Multiple Daily Injections (MDI) therapy — Injecting insulin as per participant's need.
  Arms: Group B: MDI, then Accu-Chek® Solo

SUMMARY:
This interventional device study aims to compare mainly standard Multiple Daily Injection (MDI) therapy vs. Accu-Chek® Solo Micropump System and investigates participant satisfaction. In addition, a third arm is included to compare to only similar product on the market which is OmniPod. The third arm is for data collection purpose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 1 diabetes mellitus
* At least 6 months experience with MDI therapy
* Age ≥18 years and age ≤ 65
* Able to perform carbohydrate counting
* Clinically suitable for CSII including willingness to measure blood glucose at least 4 times per day or to use flash or real-time continuous glucose monitoring consistently
* HbA1c between 7.5% (58 millimoles per mole (mmol/mol)) and 9.0% (75 mmol/mol) (determined within the last 2 months)
* Ability and willingness to read and understand study materials (participant information, data protection and written consent form, all questionnaires etc.) and to comply with study procedures
* Ability and willingness to use investigational devices independently and respond to alarms after training and run-in phase
* Using a blood glucose (BG)-meter or real-time continuous glucose monitoring device that can be downloaded via Accu-Chek® Smart Pix or willingness to use a compatible meter that will be provided for the duration of the study

Exclusion Criteria:

* Prior insulin pump use
* Relevantly impaired hypoglycemia awareness
* History of >1 hospitalization due to severe hypoglycemia within the previous 3 months
* History of >1 hospitalization due diabetic ketoacidosis within the last 3 months
* Significant manifestation of diabetes-related late complications
* Pregnant or planning to become pregnant or breastfeeding
* Known allergic reactions to plaster adhesive
* Chronic use (therapy lasting for more than 3 months) of steroids in adrenal suppressive doses, immunosuppressive medication, or chemotherapy
* Serious or unstable chronic medical or psychological condition(s)
* Addiction to alcohol or other substance(s) of abuse as determined by the investigator
* Psychological condition rendering the participant unable to understand the nature and the scope of the study
* Plans for relocation or extensive travel
* Participation in another clinical study within 4 weeks prior to the screening visit
* Dependency on Sponsor or Investigator (e.g. co-worker or family member)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Vesper, Study Director — Hoffmann-La Roche
Locations (21):
- Austria (6):
  - VIVIT Institut am LKH Felkirch, Feldkirch
  - LKH Graz, Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Salzburger Landeskliniken - Universitätsklinikum Salzburg (SALK), Salzburg
  - Diakonissen & Wehrle Privatklinik GmbH, Standort Andräviertel, Salzburg
  - Hietzing Hospital, Vienna
- Germany (6):
  - Diabetes Klinik Bad Mergentheim GmbH, Bad Mergentheim
  - InnoDiab Forschung GmbH, Essen
  - Gemeinschaftspraxis im Altstadt-Carree, Fulda
  - Gemeinschaftspraxis Drs Bieber Kraus Nolte Vortherms, Lage
  - Diabeteszentrum am CKQ, Quakenbrück
  - Diabendo Praxiszentrum, Rostock
- Poland (3):
  - Regionalne Centrum Diabetologii - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Jagiellonian University, Krakow
  - Central Clinical Hospital of the MSWiA in Warsaw, Warsaw
- United Kingdom (6):
  - Bournemouth Diabetes and Endocrine Centre, Bournemouth
  - Wolfson Diabetes & Endocrine Clinic, Cambridge
  - Centre for Clinical Research and Innovation, Darlington
  - King's College London, Diabetes Research Group, London
  - Imperial College London, Diabetes, Endocrinology and Metabolism Division, London
  - Manchester Royal Infirmary, University Hospital, Manchester

REFERENCES:
- [Derived] Barnard-Kelly K, Thienel F, Mader JK, Oliver N, Franek E, Vesper I, Dagenbach N, Vogt G, Etter T, Kunsting T. A Three-Arm Randomized Controlled Study Comparing Patient-Reported Outcomes in People With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion or Multiple Daily Injections. J Diabetes Sci Technol. 2025 Sep;19(5):1310-1316. doi: 10.1177/19322968241234055. Epub 2024 Mar 8. PMID 38456441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in 4 countries.
Pre-assignment Details: A total of 187 participants were screened into this study, of whom 6 participants were screen failures meaning that a total of 181 participants were randomised into this study.
Period: Overall Study
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Started (Full Analysis Set) | 62 | 61 | 58
Participants at End of Parallel Phase (Week 26) | 55 | 58 | 52
Completed (Week 39 (End of Solo Phase)) | 53 | 49 | 40
Not Completed | 9 | 12 | 18
Not completed — Withdrawal by Subject | 4 | 7 | 6
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Personal Reasons | 1 | 0 | 1
Not completed — Covid-19 | 1 | 4 | 3
Not completed — Multiple Reasons | 0 | 1 | 1
Not completed — Eligibility Criteria | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo | Total
Number analyzed (Participants) | 62 | 61 | 58 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (11.8) | 38.6 (10.8) | 40.6 (13.1) | 39.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 21 | 79
  Male | 33 | 32 | 37 | 102
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 59 | 60 | 56 | 175
  Asian | 1 | 1 | 1 | 3
  Other | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction: Accu-Chek® Micropump System vs. MDI, Measured by the Difference in the Diabetes Technology Questionnaire (DTQ) Total Change Score
Description: The two comparisons will be performed using a hierarchical procedure. First, the comparison between the Accu-Chek® Solo system vs. MDI will be performed and only if the corresponding Null hypothesis of no difference between both systems can be rejected, then the second comparison between Accu-Chek® Solo system and versus mylife™ OmniPod® will also be performed. The DTQ questionnaire consists of 30 questions with the individual Change Scores ranging from 1 to 5, where 1 represents 'Much worse' and 5 represents 'Much better'. The Total Change Score Range on this questionnaire is from 30 to 150 with higher scores representing lower impairment and improved outcomes.
Time Frame: 26 weeks
Population: The Full Analysis Set was defined as all eligible participants who were randomized to one of the three treatment arms.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 61
Scores on a Scale | 105.9 (2.66) | 94.8 (2.63)

2. Primary Outcome: Treatment Satisfaction: Accu-Chek® Micropump System vs. Mylife™ OmniPod®, Measured by the Difference in the Diabetes Technology Questionnaire (DTQ) Total Change Score
Description: as for outcome 1
Time Frame: 26 weeks
Population: The Full Analysis Set was defined as all eligible participants who were randomized to one of the three treatment arms.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Group A: Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 58
Scores on a Scale | 105.1 (3.04) | 108.7 (2.85)

3. Secondary Outcome: Diabetes-Related Emotional Distress Assessed by Problem Areas in Diabetes Scale (PAID)-5
Description: The PAID-5 questionnaire consisted of 5 questions with answers ranging from 0 (not a problem) to 4 (serious problem). The total score was calculated as the sum of the individual questions, resulting in a number between 0 and 20 where lower scores represented lower distress.
Time Frame: Week 26 up to Week 39
Population: The Full Analysis Set was defined as all eligible participants who were randomized to one of the three treatment arms.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 61 | 58
Scores on a Scale
  Week 26 | 7.0 (4.7) | 7.8 (4.3) | 5.3 (3.5)
  Week 39 | 6.3 (4.2) | 7.1 (4.5) | 5.8 (3.8)

4. Secondary Outcome: Device Satisfaction and Treatment Preference
Description: Device Satisfaction and Treatment Preference was the main focus of part 2 questions of the DTQ. This part of the DTQ questionnaire consisted of individual sections with 9 questions each for the Blood Glucose Meter and Insulin Pump. Individual scores ranged from 1 (terrible) to 5 (excellent). Thus, the resulting sum score ranged from 9 to 45 for each type of device.
Time Frame: Baseline up to Week 39
Population: The Full Analysis Set was defined as all eligible participants who were randomized to one of the three treatment arms. Data presented below is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 61 | 58
Scores on a Scale
  Screening (Blood Glucose Meter): number analyzed (Participants) | 60 | 56 | 58
  Screening (Blood Glucose Meter) | 35.3 (5.7) | 33.8 (5.4) | 35.7 (5.0)
  Week 13 (Blood Glucose Meter) | 34.9 (6.1) | 34.0 (5.6) | 34.9 (5.5)
  Week 26 (Blood Glucose Meter) | 34.3 (6.1) | 33.8 (5.1) | 34.9 (6.1)
  Week 39 (Blood Glucose Meter) | 34.7 (7.3) | 34.5 (5.8) | 34.8 (5.8)
  Week 13 (Insulin Pump): number analyzed (Participants) | 58 | 0 | 53
  Week 13 (Insulin Pump) | 32.7 (7.3) |  | 35.3 (4.9)
  Week 26 (Insulin Pump): number analyzed (Participants) | 60 | 0 | 53
  Week 26 (Insulin Pump) | 33.4 (6.6) |  | 35.3 (5.1)
  Week 39 (Insulin Pump): number analyzed (Participants) | 60 | 54 | 53
  Week 39 (Insulin Pump) | 33.4 (6.9) | 33.8 (6.3) | 31.0 (7.0)

5. Secondary Outcome: Therapy Success Confirmed by Glycated Hemoglobin (Hb1Ac) Levels
Description: Change in Glycated Haemoglobin (HbA1c) Levels from Baseline to Week 39
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 60 | 60 | 53
Percentage
  HbA1c at Baseline: number analyzed (Participants) | 59 | 60 | 53
  HbA1c at Baseline | 8.0 (0.6) | 8.0 (0.5) | 8.0 (0.6)
  HbA1c after 13 weeks | 7.8 (0.8) | 8.0 (0.6) | 7.9 (0.9)
  HbA1c after 26 weeks | 7.9 (0.9) | 8.2 (0.7) | 7.9 (0.9)
  HbA1c after 39 weeks | 7.8 (0.9) | 8.2 (1.1) | 8.1 (0.9)

6. Secondary Outcome: Therapy Success Indicated by Change in Body Mass Index (BMI)
Description: This outcome measure represents one reported value calculated by combining weight and height to report BMI in kg/m^2. Change in BMI from Baseline to Week 39.
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 60 | 60 | 53
kg/m^2
  Baseline | 25.4 (3.5) | 27.1 (4.7) | 27.0 (5.2)
  Week 13 | 25.3 (3.5) | 27.1 (4.7) | 27.0 (5.2)
  Week 26 | 25.4 (3.5) | 27.3 (5.0) | 27.3 (5.0)
  Week 39 | 25.7 (3.4) | 27.4 (5.0) | 27.3 (5.2)

7. Secondary Outcome: Therapy Success Indicated by Change in Weight
Description: Change in Weight from Baseline to Week 39
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 60 | 60 | 53
kg
  Baseline | 77.2 (14.1) | 81.7 (17.7) | 83.4 (18.1)
  Week 13: number analyzed (Participants) | 57 | 58 | 52
  Week 13 | 77.6 (14.3) | 82.3 (18.0) | 83.8 (17.2)
  Week 26: number analyzed (Participants) | 55 | 58 | 52
  Week 26 | 78.4 (14.9) | 82.2 (18.2) | 84.3 (17.4)
  Week 39: number analyzed (Participants) | 55 | 52 | 48
  Week 39 | 78.8 (14.6) | 82.4 (18.2) | 81.8 (17.1)

8. Secondary Outcome: Change in Glycemic Index
Description: Change in Glycemic Index from Baseline to Week 39
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 40 | 41 | 33
mg/dL
  Baseline to Week 13: number analyzed (Participants) | 31 | 30 | 22
  Baseline to Week 13 | 77.0 (15.0) | 71.7 (15.6) | 68.1 (10.2)
  Week 13 to Week 26: number analyzed (Participants) | 33 | 28 | 27
  Week 13 to Week 26 | 75.0 (21.6) | 70.2 (13.1) | 68.9 (10.0)
  Week 26 to Week 39 | 75.0 (17.0) | 73.9 (15.2) | 77.1 (15.2)

9. Secondary Outcome: Number of Participants With Therapy Parameters Indicated by Commencement of Continuous Subcutaneous Insulin Infusion (CSII)
Description: Continuous Subcutaneous Insulin Infusion (CSII) therapy is also referred to as Insulin Pump Therapy. Presented below, are the Number of Participants for whom certain indications e.g. HbA1c goals not met, resulted in commencement of CSII therapy.
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 61 | 58
Participants
  HbA1c goals not met | 62 | 61 | 56
  Participant wish | 47 | 45 | 32
  Frequent hypoglycemia | 9 | 9 | 13
  Dawn phenomenon | 3 | 2 | 2
  Glycemic variability | 1 | 3 | 2
  Shift working | 1 | 0 | 1

10. Secondary Outcome: Change in Therapy Parameters Based on Type of Insulin Used
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Number; unit: U/kg
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 61 | 58
U/kg
  Short Acting Insulin: Insulin aspart (Screening) | 37 | 30 | 39
  Short Acting Insulin: Insulin glulisine (Screening) | 2 | 9 | 2
  Short Acting Insulin: Insulin lispro (Screening) | 21 | 22 | 17
  Short Acting Insulin: Regular human insulin (Screening) | 2 | 0 | 0
  Long Acting Insulin: Insulatard (Screening) | 1 | 1 | 0
  Long Acting Insulin: Insulin degludec (Screening) | 9 | 9 | 13
  Long Acting Insulin: Insulin detemir (Screening) | 10 | 12 | 13
  Long Acting Insulin: Insulin glargine (Screening) | 42 | 38 | 32
  Long Acting Insulin: Protaphane (Screening) | 0 | 1 | 0
  Short Acting Insulin: Insulin aspart (Week 13): number analyzed (Participants) | 56 | 25 | 52
  Short Acting Insulin: Insulin aspart (Week 13) | 34 | 11 | 32
  Short Acting Insulin: Insulin glulisine (Week 13): number analyzed (Participants) | 56 | 25 | 52
  Short Acting Insulin: Insulin glulisine (Week 13) | 2 | 5 | 0
  Short Acting Insulin: Insulin lispro (Week 13): number analyzed (Participants) | 56 | 25 | 52
  Short Acting Insulin: Insulin lispro (Week 13) | 20 | 9 | 20
  Long Acting Insulin: Insulin degludec (Week 13): number analyzed (Participants) | 1 | 25 | 0
  Long Acting Insulin: Insulin degludec (Week 13) | 0 | 3 |
  Long Acting Insulin: Insulin detemir (Week 13): number analyzed (Participants) | 1 | 25 | 0
  Long Acting Insulin: Insulin detemir (Week 13) | 0 | 8 |
  Long Acting Insulin: Insulin glargine (Week 13): number analyzed (Participants) | 1 | 25 | 0
  Long Acting Insulin: Insulin glargine (Week 13) | 1 | 14 |
  Short Acting Insulin: Insulin aspart (Week 26): number analyzed (Participants) | 55 | 44 | 52
  Short Acting Insulin: Insulin aspart (Week 26) | 34 | 20 | 32
  Short Acting Insulin: Insulin glulisine (Week 26): number analyzed (Participants) | 55 | 44 | 52
  Short Acting Insulin: Insulin glulisine (Week 26) | 2 | 7 | 0
  Short Acting Insulin: Insulin lispro (Week 26): number analyzed (Participants) | 55 | 44 | 52
  Short Acting Insulin: Insulin lispro (Week 26) | 19 | 16 | 20
  Short Acting Insulin: NovoRapid (Week 26): number analyzed (Participants) | 55 | 44 | 52
  Short Acting Insulin: NovoRapid (Week 26) | 0 | 1 | 0
  Long Acting Insulin: Insulin degludec (Week 26): number analyzed (Participants) | 1 | 44 | 0
  Long Acting Insulin: Insulin degludec (Week 26) | 0 | 10 |
  Long Acting Insulin: Insulin detemir (Week 26): number analyzed (Participants) | 1 | 44 | 0
  Long Acting Insulin: Insulin detemir (Week 26) | 0 | 9 |
  Long Acting Insulin: Insulin glargine (Week 26): number analyzed (Participants) | 1 | 44 | 0
  Long Acting Insulin: Insulin glargine (Week 26) | 1 | 25 |
  Short Acting Insulin: Insulin aspart (Week 39): number analyzed (Participants) | 60 | 57 | 53
  Short Acting Insulin: Insulin aspart (Week 39) | 36 | 27 | 32
  Short Acting Insulin: Insulin glulisine (Week 39): number analyzed (Participants) | 60 | 57 | 53
  Short Acting Insulin: Insulin glulisine (Week 39) | 2 | 8 | 0
  Short Acting Insulin: Insulin lispro (Week 39): number analyzed (Participants) | 60 | 57 | 53
  Short Acting Insulin: Insulin lispro (Week 39) | 22 | 22 | 21
  Long Acting Insulin: Insulin degludec (Week 39): number analyzed (Participants) | 4 | 7 | 4
  Long Acting Insulin: Insulin degludec (Week 39) | 3 | 1 | 0
  Long Acting Insulin: Insulin detemir (Week 39): number analyzed (Participants) | 4 | 7 | 4
  Long Acting Insulin: Insulin detemir (Week 39) | 1 | 3 | 2
  Long Acting Insulin: Insulin glargine (Week 39): number analyzed (Participants) | 4 | 7 | 4
  Long Acting Insulin: Insulin glargine (Week 39) | 0 | 3 | 2

11. Secondary Outcome: Change in Therapy Parameters Indicated by Total Daily Insulin Dose (TDD)
Description: Total Daily Insulin Dose at Baseline compared to dose at Week 39
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 60 | 60 | 53
U/kg
  Screening | 0.7 (0.2) | 0.6 (0.2) | 0.7 (0.2)
  Week 13: number analyzed (Participants) | 57 | 58 | 52
  Week 13 | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2)
  Week 26: number analyzed (Participants) | 55 | 58 | 52
  Week 26 | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2)
  Week 39: number analyzed (Participants) | 55 | 52 | 48
  Week 39 | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2)

12. Secondary Outcome: Change in Therapy Parameters Indicated by Total Daily Basal Insulin Dose (TBD)
Description: Total Daily Basal Insulin Dose at Baseline compared to dose at Week 39
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 60 | 60 | 53
U/kg
  Screening | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.1)
  Week 13: number analyzed (Participants) | 57 | 58 | 52
  Week 13 | 0.3 (0.1) | 0.3 (0.1) | 0.2 (0.1)
  Week 26: number analyzed (Participants) | 55 | 58 | 52
  Week 26 | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.1)
  Week 39: number analyzed (Participants) | 55 | 52 | 48
  Week 39 | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.1)

13. Secondary Outcome: Change in Therapy Parameters Based on Average Number of Self Monitoring of Blood Glucose (SMBGs) Per Day
Description: Average Number of Self Monitoring of Blood Glucose (SMBGs) per day from Baseline up to Week 39
Time Frame: Baseline up to Week 39
Population: The Full Analysis Set was defined as all eligible participants who were randomized to one of the three treatment arms. Please note that for this Outcome Measure, incomplete SMBG data was collected which meant that data for Weeks 13, 26 and 39 could not be calculated.
Measure: Mean (Standard Deviation); unit: SMBGs per day
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 62 | 61 | 58
SMBGs per day | 3.2 (3.0) | 3.4 (3.8) | 2.5 (3.1)

14. Secondary Outcome: Percentage of Time Spent in Hypoglycaemic Blood Glucose (BG) Ranges
Description: Change in Frequency of Hypoglycaemic Events are reported below as the percentage of time spent in hypoglycaemic blood glucose (BG) ranges.
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of Time Spent
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 48 | 33 | 38
Percentage of Time Spent
  <54 mg/dL (Baseline to Week 13): number analyzed (Participants) | 48 | 27 | 38
  <54 mg/dL (Baseline to Week 13) | 3.0 (7.5) | 1.6 (2.1) | 1.1 (1.9)
  <54 mg/dL (Week 13 to Week 26): number analyzed (Participants) | 43 | 23 | 24
  <54 mg/dL (Week 13 to Week 26) | 1.8 (3.5) | 1.6 (1.9) | 0.9 (2.1)
  <54 mg/dL (Week 26 to Week 39): number analyzed (Participants) | 34 | 33 | 23
  <54 mg/dL (Week 26 to Week 39) | 1.7 (2.2) | 0.8 (1.1) | 1.1 (2.9)
  >=54 and <70 mg/dL (Baseline to Week 13): number analyzed (Participants) | 48 | 27 | 38
  >=54 and <70 mg/dL (Baseline to Week 13) | 5.8 (6.5) | 4.5 (3.0) | 3.1 (5.6)
  >=54 and <70 mg/dL (Week 13 to Week 26): number analyzed (Participants) | 43 | 23 | 24
  >=54 and <70 mg/dL (Week 13 to Week 26) | 4.9 (6.2) | 4.2 (4.2) | 3.2 (4.5)
  >=54 and <70 mg/dL (Week 26 to Week 39): number analyzed (Participants) | 34 | 33 | 23
  >=54 and <70 mg/dL (Week 26 to Week 39) | 5.6 (5.5) | 3.0 (3.1) | 1.4 (2.0)
  <70 mg/dL (Baseline to Week 13): number analyzed (Participants) | 48 | 27 | 38
  <70 mg/dL (Baseline to Week 13) | 8.8 (9.4) | 6.1 (4.7) | 4.2 (6.2)
  <70 mg/dL (Week 13 to Week 26): number analyzed (Participants) | 43 | 23 | 24
  <70 mg/dL (Week 13 to Week 26) | 6.7 (8.8) | 5.8 (5.1) | 4.1 (4.8)
  <70 mg/dL (Week 26 to Week 39): number analyzed (Participants) | 34 | 33 | 23
  <70 mg/dL (Week 26 to Week 39) | 7.3 (6.8) | 3.8 (3.7) | 2.5 (3.5)

15. Secondary Outcome: Percentage of Time Spent in Hyperglycaemic Blood Glucose (BG) Ranges
Description: Change in Frequency of Hyperglycaemic Events are reported below as the percentage of time spent in hyperglycaemic blood glucose (BG) ranges.
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of Time Spent
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 48 | 33 | 38
Percentage of Time Spent
  >180 to <250 mg/dL (Baseline to Week 13): number analyzed (Participants) | 48 | 27 | 38
  >180 to <250 mg/dL (Baseline to Week 13) | 19.3 (11.0) | 25.9 (9.0) | 26.4 (11.4)
  >180 to <250 mg/dL (Week 13 to Week 26): number analyzed (Participants) | 43 | 23 | 24
  >180 to <250 mg/dL (Week 13 to Week 26) | 19.3 (12.6) | 25.5 (7.9) | 25.4 (12.1)
  >180 to <250 mg/dL (Week 26 to Week 39): number analyzed (Participants) | 34 | 33 | 23
  >180 to <250 mg/dL (Week 26 to Week 39) | 20.3 (8.9) | 21.6 (10.1) | 26.6 (10.5)
  >250 mg/dL (Baseline to Week 13): number analyzed (Participants) | 48 | 27 | 38
  >250 mg/dL (Baseline to Week 13) | 17.4 (10.4) | 19.5 (9.5) | 16.4 (12.4)
  >250 mg/dL (Week 13 to Week 26): number analyzed (Participants) | 43 | 23 | 24
  >250 mg/dL (Week 13 to Week 26) | 15.6 (12.5) | 18.9 (8.1) | 21.0 (15.5)
  >250 mg/dL (Week 26 to Week 39): number analyzed (Participants) | 34 | 33 | 23
  >250 mg/dL (Week 26 to Week 39) | 20.3 (19.3) | 26.8 (17.2) | 29.2 (16.7)

16. Secondary Outcome: Number of Consultations
Description: Consultations between scheduled visits, emergency and call center calls, hospitalizations and absenteeism from work/school.
Time Frame: Baseline up to Week 39
Population: Please note that this Outcome Measure was not analysed because data was not collected.
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Number of Pods/Infusion Assemblies Falling Off Prematurely
Time Frame: Baseline up to Week 39
Population: Please note that this Outcome Measure was not analysed because data was not collected.
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Average Time Spent on Infusion Assembly
Time Frame: Baseline up to Week 39
Population: Please note that this Outcome Measure was not analysed because data was not collected.
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Skin Reactions (Including Type and Intensity)
Description: Number of Participants who experienced Skin Reactions at the Insulin Pump Insertion Sites (along with their Type and Intensity) are presented below, from Baseline up to Week 39. Participants were asked to assess five different properties describing potential problems at the pump insertion site, namely "itching", "redness", "swelling", "heat" and "pain". Each of these questions could be answered with one of four alternatives, "None", "Minor", "Moderate" and "Severe".
Time Frame: Baseline up to Week 39
Population: as for outcome 4
Measure: Number; unit: Number of Participants
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 60 | 60 | 53
Number of Participants
  Baseline (Itching) (Minor Intensity) | 2 | 1 | 1
  Baseline (Itching) (Moderate Intensity) | 0 | 0 | 0
  Baseline (Itching) (Severe Intensity) | 0 | 0 | 0
  Week 13 (Itching) (Minor Intensity) | 4 | 0 | 4
  Week 13 (Itching) (Moderate Intensity) | 2 | 0 | 1
  Week 13 (Itching) (Severe Intensity) | 0 | 0 | 1
  Week 26 (Itching) (Minor Intensity) | 6 | 2 | 2
  Week 26 (Itching) (Moderate Intensity) | 0 | 0 | 5
  Week 26 (Itching) (Severe Intensity) | 0 | 0 | 0
  Week 39 (Itching) (Minor Intensity) | 5 | 8 | 3
  Week 39 (Itching) (Moderate Intensity) | 0 | 3 | 3
  Week 39 (Itching) (Severe Intensity) | 1 | 0 | 2
  Baseline (Redness) (Minor Intensity) | 1 | 3 | 3
  Baseline (Redness) (Moderate Intensity) | 0 | 0 | 0
  Baseline (Redness) (Severe Intensity) | 0 | 0 | 0
  Week 13 (Redness) (Minor Intensity) | 8 | 4 | 11
  Week 13 (Redness) (Moderate Intensity) | 2 | 0 | 5
  Week 13 (Redness) (Severe Intensity) | 0 | 0 | 0
  Week 26 (Redness) (Minor Intensity) | 15 | 3 | 9
  Week 26 (Redness) (Moderate Intensity) | 0 | 0 | 4
  Week 26 (Redness) (Severe Intensity) | 0 | 0 | 0
  Week 39 (Redness) (Minor Intensity) | 16 | 11 | 10
  Week 39 (Redness) (Moderate Intensity) | 1 | 6 | 6
  Week 39 (Redness) (Severe Intensity) | 0 | 1 | 1
  Baseline (Swelling) (Minor Intensity) | 1 | 0 | 0
  Baseline (Swelling) (Moderate Intensity) | 1 | 0 | 0
  Baseline (Swelling) (Severe Intensity) | 0 | 0 | 0
  Week 13 (Swelling) (Minor Intensity) | 3 | 1 | 7
  Week 13 (Swelling) (Moderate Intensity) | 2 | 0 | 3
  Week 13 (Swelling) (Severe Intensity) | 0 | 0 | 0
  Week 26 (Swelling) (Minor Intensity) | 5 | 0 | 3
  Week 26 (Swelling) (Moderate Intensity) | 0 | 0 | 1
  Week 26 (Swelling) (Severe Intensity) | 0 | 0 | 0
  Week 39 (Swelling) (Minor Intensity) | 2 | 1 | 6
  Week 39 (Swelling) (Moderate Intensity) | 0 | 4 | 2
  Week 39 (Swelling) (Severe Intensity) | 0 | 0 | 0
  Baseline (Heat) (Minor Intensity) | 0 | 0 | 0
  Baseline (Heat) (Moderate Intensity) | 0 | 0 | 0
  Baseline (Heat) (Severe Intensity) | 0 | 0 | 0
  Week 13 (Heat) (Minor Intensity) | 1 | 0 | 3
  Week 13 (Heat) (Moderate Intensity) | 1 | 1 | 0
  Week 13 (Heat) (Severe Intensity) | 0 | 0 | 0
  Week 26 (Heat) (Minor Intensity) | 0 | 0 | 1
  Week 26 (Heat) (Moderate Intensity) | 0 | 0 | 1
  Week 26 (Heat) (Severe Intensity) | 0 | 0 | 0
  Week 39 (Heat) (Minor Intensity) | 1 | 1 | 1
  Week 39 (Heat) (Moderate Intensity) | 0 | 1 | 0
  Week 39 (Heat) (Severe Intensity) | 0 | 1 | 0
  Baseline (Pain) (Minor Intensity) | 4 | 3 | 3
  Baseline (Pain) (Moderate Intensity) | 0 | 0 | 2
  Baseline (Pain) (Severe Intensity) | 0 | 0 | 0
  Week 13 (Pain) (Minor Intensity) | 3 | 1 | 3
  Week 13 (Pain) (Moderate Intensity) | 1 | 1 | 2
  Week 13 (Pain) (Severe Intensity) | 1 | 0 | 0
  Week 26 (Pain) (Minor Intensity) | 3 | 3 | 3
  Week 26 (Pain) (Moderate Intensity) | 1 | 0 | 2
  Week 26 (Pain) (Severe Intensity) | 0 | 0 | 0
  Week 39 (Pain) (Minor Intensity) | 3 | 4 | 4
  Week 39 (Pain) (Moderate Intensity) | 1 | 1 | 3
  Week 39 (Pain) (Severe Intensity) | 0 | 2 | 0

20. Secondary Outcome: Socio-economic Acceptance: Amount of Insulin Left in Device at Reservoir Change/Device Discard
Time Frame: Baseline up to Week 39
Population: Please note that this Outcome Measure was not analysed because data was not collected.
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Amount of Waste, Inferred by Total Material Consumption
Time Frame: Baseline up to Week 39
Population: Please note that this Outcome Measure was not analysed because data was not collected.
Arm/Group | Group A: Accu-Chek® Solo | Group B: MDI, Then Accu-Chek® Solo | Group C: Mylife™ OmniPod®, Then Accu-Chek® Solo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up until a maximum of 40 weeks.
Groups:
- Group A: Accu-Chek® Solo (Parallel Phase): Continuous subcutaneous insulin infusion (CSII) with Accu-Chek® Solo Micropump system for 26 weeks.
- Group B: MDI (Parallel Phase): Multiple daily injections (MDI) for 26 weeks.
- Group C: Mylife™ OmniPod® (Parallel Phase): Continuous subcutaneous insulin infusion (CSII) with the mylife™ OmniPod® Insulin Management system for 26 weeks.
- Group D: Groups A+B+C (Solo Phase): From Week 26 until Week 39, all Groups (A, B and C) used the Accu-Chek® Solo Micropump system for CSII therapy.
Arm/Group | Group A: Accu-Chek® Solo (Parallel Phase) | Group B: MDI (Parallel Phase) | Group C: Mylife™ OmniPod® (Parallel Phase) | Group D: Groups A+B+C (Solo Phase)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/61 | 0/58 | 0/165
Serious Adverse Events (participants affected / at risk) | 6/62 | 1/61 | 5/58 | 4/165
Other Adverse Events (participants affected / at risk) | 44/62 | 35/61 | 35/58 | 82/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Accu-Chek® Solo (Parallel Phase) (N=62) | Group B: MDI (Parallel Phase) (N=61) | Group C: Mylife™ OmniPod® (Parallel Phase) (N=58) | Group D: Groups A+B+C (Solo Phase) (N=165)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (2) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Accu-Chek® Solo (Parallel Phase) (N=62) | Group B: MDI (Parallel Phase) (N=61) | Group C: Mylife™ OmniPod® (Parallel Phase) (N=58) | Group D: Groups A+B+C (Solo Phase) (N=165)
Diabetic ketosis (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 4 (5) | 21 (31)
Hypoglycaemia (Metabolism and nutrition disorders) | 32 (743) | 28 (653) | 22 (183) | 49 (838)
Nasopharyngitis (Infections and infestations) | 5 (7) | 7 (9) | 9 (10) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT03478969/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT03478969/SAP_001.pdf